CLINICAL TRIAL: NCT02146807
Title: LASER TREATMENT OF TATTOOS WITH A DUAL WAVELENGTH PICOSECOND LASER
Brief Title: Laser Treatment of Tattoos With Pico Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IH132802
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Unwanted Tattoos
Keywords: Tattoos, Picosecond Laser, Syneron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosecond Laser System (Experimental)
  Interventions: Device: Picosecond Laser system

INTERVENTIONS:
Device: Picosecond Laser system — Picosecond Laser System for the Treatment of Unwanted Tattoos

SUMMARY:
The purpose of this study is to determine whether Pico laser is effective and safe in the treatment of unwanted tattoos.

DETAILED DESCRIPTION:
The Investigational device is a dual wavelength laser system developed for treatment of pigmented lesions and for tattoo removal. The base unit is a GentleMax Pro laser system modified to emit light at wavelengths of 532 and 1064 nm and deliver pulse energy up to 400mJ, and pulse duration of 700 ps.

A multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Has Fitzpatrick skin type I-IV
2. Has unwanted non-cosmetic tattoo(s) and wishes to undergo laser treatments to remove them
3. Is willing to consent to participate in the study
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits

Exclusion Criteria:

1. Is hypersensitive to light exposure
2. Has an active sun tan
3. Has Fitzpatrick skin type V or VI
4. Has active localized or systemic infection
5. Is taking medication(s) for which sunlight is a contraindication
6. Has a history of squamous cell carcinoma or melanoma
7. Has a history of keloid scarring
8. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment.
9. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications
10. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period
11. Is allergic to lidocaine, tetracaine or Xylocaine with epinephrine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Global percentage of tattoo clearance | 3 months post the final treatment
  Global percentage of tattoo clearance evaluated by blinded observers using post treatment photographs compared to baseline photographs.

SECONDARY OUTCOMES:
Rate of tattoo clearance | 3 months
  The average number of treatments will be determined in order to obtain 50% and 75% tattoo clearance. Rate of clearance will be assessed globally independent of tattoo color and based on individual colors.

OTHER OUTCOMES:
Number of Participants with Adverse Events | 3 months
  Adverse events will be evaluated immediately after and before each subsequent laser treatment and will be based on the incidence and severity of side effects caused by the laser treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, Study Director — Syneron Medical Ltd.
Locations (3):
- United States (3):
  - Washington Institute of Dermatologic Laser Surgery, Washington D.C., District of Columbia
  - New York Laser and Skin Care, New York, New York
  - Main Line Center for Laser Surgery, Ardmore, Pennsylvania